CLINICAL TRIAL: NCT06517940
Title: A Prospective, Observational Study in Adults With Retinitis Pigmentosa (RP)
Status: Active, not recruiting | Type: Observational
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DE101111
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis Pigmentosa. Natural history
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The natural history in individuals with severe retinitis pigmentosa (RP) is variable and there remains an unmet need to better understand disease progression in this population. The goal of this study is to determine which visual assessments individuals with RP and low visual acuity can reliably perform and to evaluate the annual decline of visual function in severe RP.

DETAILED DESCRIPTION:
This is a 12-month, single-center, prospective observational study in adults with RP. Approximately 12 subjects will be enrolled into the Observation Period.

The primary objective of this study is to determine which visual assessments RP subjects with low visual acuity can reliably perform. Other objectives are 1) to determine which visual assessments are most sensitive to annual change in RP subjects with low visual acuity, 2) to evaluate adverse events, 3) to evaluate the safety and tolerability of study assessment procedures, and 4) to evaluate the subject's experience in this study, relevance of visual assessments and patient-reported outcome measures, and perception of improvement in visual function.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age at the time of informed consent.
* Subject has a clinical diagnosis of nonsyndromic retinitis pigmentosa.
* Subject is willing to consent to genetic testing, if not already done.
* Subject has BCVA in the worse eye between hand motion and 35 Early Treatment of Diabetic Retinopathy Study (ETDRS) letter score (approximately ≤ 20/200 Snellen equivalent), inclusive.
* Subject has a central visual field diameter (ie, excluding temporal islands) of < 20 degrees in the worse eye as measured with the V4e stimulus using kinetic perimetry.

Exclusion Criteria:

* Subject has an eye disease or visual disorder other than retinitis pigmentosa that impairs visual function.
* Subject has any other eye condition, which in the opinion of the Investigator, would preclude an accurate evaluation at any time during the study.
* Subject has any clinically significant unstable medical condition or any clinically significant chronic disease that in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in the study.
* Subject has received treatment with any nonapproved, experimental, or investigational therapy in either eye (systemic, topical, intravitreal) and/or received treatment in an interventional clinical trial for an eye disease or disorder within 90 days or 5 half-lives, whichever is longer, prior to Screening or anticipates the need to receive treatment in an interventional clinical trial during their participation in this study.
* Subject has previously received cell therapy, gene augmentation therapy, genome editing therapy, or any subretinal administered therapy for an eye disease or disorder or anticipates the need for these therapies during their participation in this study.
* Subject has previously received LUXTURNA (voretigene neparvovec-rzyl) or anticipates the need for this therapy during their participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retinitis pigmentosa subjects with low visual acuity
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Reliability (test-retest variability within subjects) | 12 months
  Reliability (test-retest variability within subjects) on:
  * Total visual area (degrees squared) on kinetic perimetry using V4e stimulus (excluding temporal islands) (Time frame: 12 months)
  * Early Treatment of Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) Log of Minimum Angle of Resolution (LogMAR) equivalent (or Low Vision Test, as applicable) (Time frame: 12 months)
  * Retinal light sensitivity on Full-field Stimulus Threshold test (Time frame: 12 months)
  * Retinal sensitivity and fixation stability on microperimetry (Time frame: 12 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Mass Eye and Ear, Boston, Massachusetts, United States